CLINICAL TRIAL: NCT02732548
Title: MIRODERM™ for Complex Wounds in an Inpatient Setting
Brief Title: MIRODERM™ for Complex Wounds in an Inpatient Setting (MIRODERM CLOSure)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016001
Record Dates: First submitted 2016-03-31; First posted 2016-04-08 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Complex Wound
MeSH Terms: interventions — Negative-Pressure Wound Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPWT Only (Active Comparator): Study subjects who are randomized to the control arm will be treated with Negative Pressure Wound Therapy (NPWT) and additional standard care treatments. No cellular or acellular biological tissue scaffold will be allowed for subjects in this study arm for the first 6 weeks of the study. Subjects who are randomized to this arm and who do not experience at least a 50% surface area reduction of the study wound by the 6 week study visit will have the option to cross over into the NPWT + MIRODERM treatment arm.
  Interventions: Other: Negative Pressure Wound Therapy (NPWT); Other: Standard Care
- NPWT + MIRODERM (Experimental): Subjects in this arm will receive NPWT and standard care, plus application(s) of the MIRODERM product.
  Interventions: Other: Negative Pressure Wound Therapy (NPWT); Other: MIRODERM Application(s); Other: Standard Care

INTERVENTIONS:
Other: Negative Pressure Wound Therapy (NPWT)
Other: MIRODERM Application(s)
  Arms: NPWT + MIRODERM
Other: Standard Care — wound measurement, debridement, photography of wound, moist wound environment, infection management, nutritional support

SUMMARY:
This study is being conducted to collect data on the performance of Miromatrix Wound Matrix (MIRODERM) when used in the treatment of complex wounds in an inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Have a complex study wound which will require an autograft or delayed primary closure procedure and which may or may not include tunneling and/or undermining
* Have a study wound with a total post-debridement surface area ≥50cm2 and ≤250cm2 with no dimension >25cm, and a minimum depth of ≥0.5cm
* Have a study wound which is expected to take at least 4 weeks to reach autograft or delayed primary closure using standard care and NPWT
* Have a study wound that will be treated with NPWT regardless of study participation
* Be in an inpatient setting
* Be able and willing to sign the consent form and comply with all study visits and procedures

Exclusion Criteria:

* Be pregnant or be planning to become pregnant during the study
* Be contraindicated for NPWT (necrotic tissue with eschar present, untreated osteomyelitis, non-enteric and unexplored fistulas, malignancy in the wound, exposed vasculature, exposed nerves, exposed anastomotic site, exposed organs)
* Be immunocompromised or at risk of immunosuppression (e.g. be HIV positive, be experiencing organ rejection, be a recent, current, or anticipated chemotherapy recipient) as determined by the Investigator
* Be taking a Tumor Necrosis Factor (TNF) blocker
* Be participating in another research study
* Have a sensitivity to porcine material
* Have a life expectancy of less than 1 year
* Have a study wound which is a third degree burn wound
* Have a study wound that is infected
* Have a study wound that is a pressure ulcer/wound
* Have a study wound with sinus tract(s) leading to other open area(s)
* Have a wound that is being treated or expected to be treated with either HBOT or topical wound oxygen therapy
* Have a study wound which has been treated with a cellular and/or tissue-based product within last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects that have had an autograft or delayed primary closure procedure for the study wound by Week 6. | 6 weeks
  The primary endpoint is the proportion of subjects that have had an autograft or delayed primary closure procedure for the study wound by the 6 week visit.